CLINICAL TRIAL: NCT05250063
Title: A Multicenter, Open-Label, Phase 2 Study to Evaluate Growth and Safety of LUM-201 Following 12 Months of Daily rhGH Treatment in Children With Idiopathic Growth Hormone Deficiency Who Have Previously Completed the LUM-201-01 Trial
Brief Title: Phase 2 Study of LUM-201 in Children Who Have Previously Completed the LUM-201-01 Trial (OraGrowtH213)
Acronym: OraGrowtH213
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumos Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-201-04
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Growth Hormone Deficiency
Keywords: LUM-201; PGHD; Height; Oral
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LUM-201 (3.2 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201

INTERVENTIONS:
Drug: LUM-201 — Administered orally once daily

SUMMARY:
This is a multi-national trial. The goals of the trial are to study the growth response to LUM-201 administration in children with idiopathic growth hormone deficiency (GHD) previously treated with daily rhGH for 12 months in the LUM-201-01 trial.

DETAILED DESCRIPTION:
This trial will have one screening/baseline visit with tests to assess if subjects are eligible to start study therapy. The screening/baseline visit can coincide with the Month 12 visit in the LUM-201-01 trial. Subjects will receive the same dose of LUM-201 as a daily oral dose each morning. LUM-201 will be adjusted for body weight increments at each clinic visit, as applicable.

The trial consists of 12 months of treatment. After screening, subjects will return to the clinic for 5 visits. During four of these clinic visits, safety laboratory samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver must sign the informed consent, and the subject must sign the assent, as applicable.
* Must have previously completed 12 months of daily rhGH treatment as part of the LUM-201-01 PGHD trial.
* Is eligible for study participation as confirmed by the principal investigator (PI)

Exclusion Criteria:

* Has a medical condition that, in the opinion of the PI and/or MM, adds unwarranted risk to use of LUM-201.
* Uses any medication that, in the opinion of the PI and/or MM, can independently cause short stature or limit the response to exogenous growth factors.
* Has planned or is receiving current long-term treatment with medications known to act as substrates, inducers, or inhibitors of the cytochrome system CYP3A4 that metabolizes LUM-201

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Annualized height velocity (AHV) measured as standing height with stadiometer | Day 1 to Month 12
  Annualized Height Velocity (AHV) measured as standing height with stadiometer

SECONDARY OUTCOMES:
Incidence of adverse events in children with GHD | Day 1 to Month 12
  Number of events
GH Concentration on maintenance treatment | Day 1 to Month 12
  Serum GH concentration
Insulin-like growth factor 1 | Day 1 to Month 12
  Serum concentrations of insulin-like growth factor 1
Insulin-like growth factor binding protein 3 | Day 1 to Month 12
  Serum concentrations of insulin-like growth factor binding protein 3
Height standard deviation score (SDS) | Day 1 to Month 12
  Change in HT-SDS
Change in Weight | Day 1 to Month 12
  Change in Weight
Change in Weight-SDS | Day 1 to Month 12
  Change in Weight-SDS
Change in BMI | Day 1 to Month 12
  Change in BMI
Change in BMI SDS | Day 1 to Month 12
  Change in BMI SDS
Change in Bone Age | Month 6
  Change in bone age, measured by X-ray of left hand and wrist using Greulich & Pyle atlas
Insulin-like growth factor 1 standard deviation score (SDS) | Day 1 to Month 12
  Change in IGF-1 SDS

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - Rady Children's Hospital, San Diego, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - M Health, Fairview Pediatric Specialty Clinics- Discovery Clinic, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Virginia Health System, Charlottesville, Virginia
- Poland (3):
  - Klinika Endokrynologii i Chorob Metabolicznych, Instytut Centrum Zdrowia Matki Polki, Lodz
  - Sonomed - Centrum Medyczne, Szczecin
  - Klinika Endokrynologii i Diabetologii, Instytut "Pomnik Centrum Zdrowia Dziecka, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided